CLINICAL TRIAL: NCT03784547
Title: Real-world Patient Profile and Treatment Persistence of Ocrelizumab in Multiple Sclerosis: A Retrospective Analysis in Latin America
Brief Title: Real-world Data of Ocrelizumab in Multiple Sclerosis in LATAM
Acronym: RWD_ocre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: RWD_Ocrelizumab LATAM
Record Dates: First submitted 2018-12-13; First posted 2018-12-24 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Latin america
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple sclerosis patients: multiple sclerosis patients receiving ocrelizumab 600 mg endovenous every 6 months
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — already described
  Other Names: no other

SUMMARY:
It has been almost 25 years since the publication of the pivotal trial results for the first disease-modifying therapy (DMT) for RRMS. Currently disease modifying therapies (DMTs) for MS approved by the European Medicine Agency (EMA) and Food and Drug Administration (FDA) include interferon beta (IFNβ) 1-a and 1-b, glatiramer acetate (GA), mitoxantrone, natalizumab, fingolimod, teriflunomide, dimethyl fumarate, alemtuzumab, daclizumab and ocrelizumab. Despite evidence about ocrelizumab exist in many patients from eurpe and North America, scarce real world evidence exists about epidemiolofcal aspects of patients that used ocrelizumab in Latin America.

The aim of this study is therefore to evaluate patient profiles and persistence to treatment during follow up in a retrospective study of patients who had been prescribed ocrelizumab for the treatment of MS in Latin America (LATAM). The investigators will include MS patients that received ocrelizumab in Latin America and describe epidemiological aspects and persistence to treatment during the last 12 months.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic inflammatory disease of the CNS that leads to focal plaques of primary demyelination and diffuse neurodegeneration in the grey and white matter of the brain and spinal cord 1. In most patients, the disease starts with a relapsing-remitting course (RRMS), which is followed several years by a secondary progressive phase (SPMS). Patients with primary progressive disease (PPMS) miss the relapsing and remitting stage and start with uninterrupted progression from disease onset 1-3.

It has been almost 25 years since the publication of the pivotal trial results for the first disease-modifying therapy (DMT) for RRMS 4. Currently disease modifying therapies (DMTs) for MS approved by the European Medicine Agency (EMA) and Food and Drug Administration (FDA) include interferon beta (IFNβ) 1-a and 1-b, glatiramer acetate (GA), mitoxantrone, natalizumab, fingolimod, teriflunomide, dimethyl fumarate, alemtuzumab, daclizumab and ocrelizumab 5-7.

Ocrelizumab was approved in March 2017 for the treatment of relapsing or primary progressive MS 8. A phase II trial established 600 mg intravenously every 6 months as the preferred dosing schedule. Two phase III trials evaluated the efficacy of ocrelizumab in patients with relapsing remitting MS, and individual and pooled analysis demonstrated a significant reduction in annualized relapse rate (P < 0.001 pooled), disability progression at 12 weeks ( P < 0.001 pooled), and gadolinium-enhancing lesions on magnetic resonance imaging (MRI; P < 0.001) 8. Patients with PPMS were evaluated in a third phase III trial, which showed a significant decrease in disease progression at 12 weeks ( P = 0.03) and volume of T2-weighted lesions on MRI ( P < 0.001) 8. As with other monoclonal antibodies, adverse effects seen with ocrelizumab were primarily infusion-related reactions and infection8. Despite much information exists about efficacy and safety of ocrelizumab in phase III clinical trials, scarce evidence exists regarding real world patients profile and safety.

The aim of this study is therefore to evaluate patient profiles and persistence to treatment during follow up in a retrospective study of patients who had been prescribed ocrelizumab for the treatment of MS in Latin America (LATAM)

Methods

Verbal/written consent from patient only if any site's Ethic Committee requests it.

Centers involved in the study will be from Mexico, Chile, Argentina Number of centers & patients Two centers in Argentina, two centers in Chile, and two centers in Mexico. Total: 6 centers and Approx 80 patients.

Study overview Patients that accept to participate and fulfill all inclusion criteria and none exclusion criteria will be included. All information will be extracted from the medical charts Data Source Information related to the study population will be extracted from the patient medical chart review (secondary data use) and will cover a period up to protocol regulatory approval. Patient identity will be coded and anonymized in the study data base so only each investigator will know the identity of each patient. Local legislation regarding patient data protection will be followed strictly in this study. All study data will be entered in a predefined electronic Case Report Form (CRF).

This is an NIS involving the use of secondary data and the reporting of adverse reactions in the form of ICSRs is not required. The study will not extract safety information.

Storage and data analysis

Once the patient is identified and consented to participate (if needed based on local regulatory aspects), data from patient's chart will be transferred into the specifically designed platform. The platform on which variables will be transferred, will be on a web platform with restricted access by user and password specific to each researcher. When sharing the data, it will be anonymized and only data related to the demographics and clinic will be accessible, and patient data such as name, surname and ID will not be visible to analysts if it is loaded.

Data protection

The regulatory requirements and protection of personal data must be completed according to the regulations corresponding to each participant.

Each researcher in the study should explain in detail to each potential participant the record consists. Every patient who wishes to participate in the project must consent, according to each regulation, authorizing that their information, codified and anonymized, be shared with other records for analysis and communication.

An institutional ethics committee must approve the registration or declare that it is exempt from the need for approval as well as its informed consent (IC).

The data will be uploaded by the physician of each participating center. The different variables will be obtained from the daily clinical practice of each professional.

Patient Confidentiality As mentioned in the previous point, the patient's name, address, date of birth, ID or telephone number will only be left in the personal registry and at the moment of sharing the registration to the central registry will not be entered. The records will then be identified by a unique code generated by the initials of the IP and the registration number of that patient.

Each registry should include baseline clinical and demographic data as well as the study project data.

At all times, the protection of the patient's identity and data will be observed in accordance with the legal regulations in force national law of protection of personal data 25.326 (Habeas Data), in accordance with the international legislation on registration of diseases and protection of personal data and private, according to the 18th World Medical Assembly of Helsinki (1964) when applicable. The right to non-participation in the study will be respected always without this implying in any case any type of discrimination, differential treatment or mistreatment towards the patient.

This is a retrospective observational study, which does not plan any type of intervention or differential treatment in patients included or excluded.

Statistical analysis plan This is descriptive study and sample size is not based on statistical considerations. A descriptive analysis is the main objective of the study regarding demographic, clinical aspects, disease activity and persistence to treatment of patients that received ocrelizumab to treat their MS disease.

ELIGIBILITY:
Inclusion Criteria:

- multiple sclerosis patients that received ocrelizumab

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must meet the following inclusion criteria:
  MS patients who received ocrelizumab to treat their disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients discontinuing the treatment with ocrelizumab in the last 12 months after inclusion | 12 months
  To describe the number of patients that discontinue the use of ocrelizumab during the last 12 months
Multiple sclerosis phenotype | 12 months
  to describe the MS phenotype of patients that received ocrelizumab in LATAM

SECONDARY OUTCOMES:
Gender | 12 months
  to describe the gender of patients that received ocrelizumab in LATAM
Age at study entry | 12 months
  To describe the age of patients that received ocrelizumab at study entry

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Juan Ignacio Rojas, Buenos Aires
  - Edgard Carnero, Buenos Aires

IPD SHARING:
Plan to Share IPD: No